CLINICAL TRIAL: NCT05401942
Title: Real-time Tele-monitoring Versus Routine Monitoring of Breast Cancer Patients Receiving Adjuvant Systemic Therapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 261\2021
Record Dates: First submitted 2022-03-12; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine monitoring (No Intervention): patients with breast cancer who will receive adjuvant treatment and will be followed up during treatment with routine visits.
- Tele-monitoring through mobile application (Active Comparator): Patients with breast cancer who will receive adjuvant therapy and will be followed up during treatment through tele-monitoring with mobile application and CTCAE checklist for PRO.
  Interventions: Other: Tele-monitoring through mobile application

INTERVENTIONS:
Other: Tele-monitoring through mobile application — Tele-monitoring of Patient reported outcomes
  Arms: Tele-monitoring through mobile application

SUMMARY:
Patients with breast cancer receiving systemic therapy have a variety of symptoms.

In cancer patients receiving chemotherapy and targeted therapy, it is common to report symptoms to physicians before each cycle of systemic therapy and planning maintenance and treatment applications accordingly. Nowadays tele-monitoring of patient reported outcomes using mobile applications is used widely.

These applications provide many advantages to the patient, physicians, and health care system because patients report the symptoms experienced and helps contribute to the quick management of the symptoms and improve the adherence to treatment, decrease the frequency of dose delays and dose reduction of their treatment.

DETAILED DESCRIPTION:
In Egypt, breast cancer is the most frequent malignancy among Egyptian women, accounting for 38.8% of cancers in this population, with the expected number of breast cancer cases nearly 22, 700 in 2020 and forecasted to be approximately 46, 000 in 2050.It is found that the breast cancer mortality rate is around 11%, being the second cause of cancer-related mortality after hepatocellular carcinoma.

Systemic therapy including chemotherapy and antiHER2 drugs are frequently utilized in the adjuvant setting in the treatment of breast cancer as Anthracycline-based chemotherapy (AC, FEC, FAC Protocols containing Doxorubicin, Epirubicin, fluorouracil and cyclophosphamide), which may lead to cardiac side effects, taxanes (Paclitaxel and Docetaxel) which may lead to GIT Problems and peripheral neuropathy. The addition of trastuzumab to a sequential anthracycline/cyclophosphamide-taxane regimen was linked to a 3% risk of cardiac toxicity, whereas trastuzumab in conjunction with non-anthracycline regimens (e.g. carboplatin/docetaxel) was linked to lower rates of cardiac toxicity.

These drugs may result in a variety of symptoms to develop, it is critical to measure, prevent and control them. Patient-reported outcomes (PROs) are becoming more popular as a way to quantify symptoms and health-related quality of life in cancer care. PROs are useful to capture the patient's perspective on their care and treatment, and they are intended to supplement traditional clinical outcomes and toxicity reported by physicians such as survival and toxicity assessment.

Tele-monitoring is crucial in patients' follow-up as it will improve patients' adherence to treatment, decrease the frequency in dose reduction and dose delay. This will be accomplished by using tele-monitoring in reporting and managing patient reported outcomes from chemotherapy using PRO- CTCAE Checklist, version 1 to assess the grade and severity of symptoms reported by patients throughout the course of adjuvant chemotherapy with early management compared to the routine monitoring done in the regular clinic visits. In order to avoid the complications, symptoms should be diagnosed early and symptom referral for management should be advised and offered with evidence-based approaches. For this purpose, symptom reporting has recently been using mobile applications.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-III breast cancer under adjuvant intravenous chemotherapy with or without targeted therapy.
2. Able to provide a written informed consent .
3. Must have an internet access.

Exclusion Criteria:

1. Presence of other malignancies whether in the past or simultaneously.
2. Male cancer patients.
3. Clinical diagnosis of Alzheimer's disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients
Enrollment: 150 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of frequency and severity of symptoms using real-time tele-monitoring versus routine symptom monitoring. | 2 years
  To compare between grade of side effects of treatment between both arms through CTCAE checklist for patient reported outcomes.

SECONDARY OUTCOMES:
● Comparison of adherence to treatment between both groups. | 3 years
  to compare the tolerability for treatment between both arms through assessment of the percentage of dose delay in both groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozturk ES, Kutluturkan S. The Effect of the Mobile Application-Based Symptom Monitoring Process on the Symptom Control and Quality of Life in Breast Cancer Patients. Semin Oncol Nurs. 2021 Jun;37(3):151161. doi: 10.1016/j.soncn.2021.151161. Epub 2021 Jun 2. PMID 34088557